CLINICAL TRIAL: NCT02246699
Title: A Study to Evaluate the Efficacy and the Safety of a Fungal Chitosan on the Body Weight Reduction in Overweight and Obesity Volunteers: a Randomized, Double-blind, Parallel Groups and Placebo Controlled Clinical Trial.
Brief Title: Efficacy and Safety of a Fungal Chitosan on the Body Weight Reduction in Overweight and Obesity Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kitozyme (Industry)
Collaborators: Naturalpha (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-041; ID-RCB Number : 2014-A01026-41 (Other: ANSM)
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Overweight and Obese Volunteers.
Keywords: obesity; overweight; chitosan; fungal chitosan; weight management
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KiOnutrime®-Cs (Experimental): The product is presented as a capsule containing chitosan as ingredient supporting the activity.
  Interventions: Device: KiOnutrime®-Cs
- Placebo (Placebo Comparator): Placebo is presented as a capsule containing inactive ingredients.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: KiOnutrime®-Cs — The product will be taken orally within 15 minutes before main meals (breakfast, lunch and dinner) with a large glass of water. Subjects will have to take 2 capsules of 500mg, 3 times per day.
  Arms: KiOnutrime®-Cs
Other: Placebo — The product will be taken orally within 15 minutes before main meals (breakfast, lunch and dinner) with a large glass of water. Subjects will have to take 2 capsules, 3 times per day.
  Arms: Placebo

SUMMARY:
The prevalence of overweight and obesity is getting more and more important in developed as well as in emerging countries. It can be defined according to the degree of fat storage by measurement of fat mass.

No clinical studies have been conducted so far for that intended use on KiOnutrime®-Cs, a fungal chitosan from the mycelium of non-genetically modified Aspergillus niger. KiOnutrime®-Cs has been recognized as substantially equivalent to animal chitosan.

The purpose of this clinical trial is to determine if KiOnutrime®-Cs-containing medical device, which is a CE-marked medical device manufactured by KitoZyme, has an effect on body weight reduction after 3 months of intake in overweight and obese men and women. Furthermore, effects on anthropometric measurements, body fat mass percentage, serum lipids and safety parameters will be investigated.

DETAILED DESCRIPTION:
The study duration per subject will be 3 months and 1 week maximum. Subjects will be screened at visit V1 and will start a 1-week run-in period, during which subjects will ingest 2 capsules of placebo 3 times a day.

The subjects will then be randomized to receive the investigational medical device or placebo (1:1) for a 3 months product intake period.

ELIGIBILITY:
Inclusion Criteria:

* Males and females volunteers, able to read and write.
* Subject with 25 ≤ Body Mass Index ≤ 35 kg/m².
* Subject with a good physical condition based on the subject's interview and the clinical exam performed by the Investigator.
* Subject with stable body weight (< 5% variation) within the last 3 months prior to screening (based on interview).
* Written informed consent provided prior to screening, after receiving and understanding the subject information.
* Subject willing to lose weight.
* Subject accepting to follow diet and lifestyle instructions throughout the study.
* Subject willing to take study capsules three times a day for 3 months and 1 week and undergo other study-related procedures.
* Registered with the French Social Security, in agreement with the French law on biomedical experimentation.

Exclusion Criteria:

* Smoker or former smoker having stopped within 2 months prior to screening visit.
* Subject with a history of alcohol or drug abuse.
* Subject with physical activity more than 3 hours per week.
* Subject with any sensitivity or allergy to any of the products used within this clinical trial.
* Subject with history of eating disorder (anorexia nervosa, bulimia nervosa).
* Subject having used weight reduction treatments or products during the last 3 months prior to screening visit.
* Subject with significant gastrointestinal disease (e.g. coeliac disease, pancreatitis), signs of intestinal obstruction or medical history of constipation.
* Intake of chronic medication which could interfere with study parameters (weight, appetite, satiety, lipid blood levels, glycemia, gastrointestinal function), having an effect on digestion or absorption of nutrients, excepted oestroprogestative or progestative contraception started at least three months before the screening visit.
* Female subject planning a pregnancy, pregnant or breastfeeding.
* Female subject without efficient contraceptive method.
* Subject with history of bariatric surgery.
* Subject with known systemic disease such as cancer, human immunodeficiency virus (HIV) seropositivity.
* Subject with type 1 or type 2 diabetes mellitus.
* Subject with history of significant medical or surgical event requiring hospitalization during the 3 months prior the screening visit.
* Subject having, had or scheduling to have an exam that uses barium, a radioisotope injection, or oral or intravenous contrast material within 2 weeks prior screening visit and during the study.
* Participation to any other clinical trial simultaneously and/or within 1 month prior the screening visit.
* Subject who has donated blood or blood products within the previous month prior to screening or who plans to donate blood or blood products at any time during the trial and in the 3 months following the end of the study.
* Subject judged unlikely to comply with study product intake (screening compliance < 80%) and with diet and lifestyle instructions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Body weight | 0 ; 30 ; 60 ; 90 days
  Comparison of the reduction of body weight, from baseline (randomization visit) to end-point (3 months of treatment), between KiOnutrime®-Cs and placebo arms.

SECONDARY OUTCOMES:
Anthropometric measurements | 0 ; 30 ; 60 ; 90 days
  Mean changes from baseline (randomization visit) to end-point (3 months of treatment) in anthropometric measurements (Body Mass Index, waist, hip and thigh circumferences) between KiOnutrime®-Cs and placebo.
Body fat mass | 0 - 90 days
  Mean changes from baseline (randomization visit) to end-point (3 months of treatment) in body fat mass percentage (fat mass, bone mass and lean mass measured by Dual-energy X-ray absorptiometry) between KiOnutrime®-Cs and placebo.
Hunger and satiety sensation | -7 ; 0 ; 30 ; 60 ; 90 days
  Mean changes from baseline (randomization visit) to end-point (3 months of treatment) in hunger and satiety sensation via Visual Analog Scales measures between KiOnutrime®-Cs and placebo.
Serum lipids | 0 - 90 days
  Mean changes from baseline (randomization visit) to end-point (3 months of treatment) in serum lipids (triglycerides and cholesterol) between KiOnutrime®-Cs and placebo.
Blood pressure | 0 ; 30 ; 60 ; 90 days
  Mean changes from baseline (randomization visit) to end-point (3 months of treatment) in systolic and diastolic blood pressure between KiOnutrime®-Cs and placebo.
Electrolytic measurements and fat-soluble vitamins | 0 - 90 days
  Mean changes from baseline (randomization visit) to end-point (3 months of treatment) in electrolytic measurements (Calcium, Magnesium, Sodium, Potassium) and fat-soluble vitamins (A, D, E) in plasma between KiOnutrime®-Cs and placebo.
Gastrointestinal tolerance | -7 ; 0 ; 30 ; 60 ; 90 days
  Evaluation of the gastrointestinal tolerance of KiOnutrime®-Cs with a questionnaire at baseline (randomization visit), 30 days, 60 days and 90 days compared to placebo.
Safety blood parameters | 0 - 90 days
  Evaluation of the safety of KiOnutrime®-Cs through safety blood parameters measurements (urea, creatinine, glucose, Aspartate Aminotransferase and Alanine Aminotransferase).
Adverse events | Study duration
  Evaluation of the safety of KiOnutrime®-Cs through adverse events recording.
Physical Activity score | -7 ; 0 ; 30 ; 60 ; 90 days
  Mean changes from baseline (randomization visit) to end-point (3 months of treatment) in Physical Activity score (via Physical activity questionnaire).
Food recording | 0 ; 30 ; 60 ; 90 days
  Estimation of total intake of food energy (calories), nutrients, and non-nutrient food components from foods and beverages that were consumed during a 3 days period prior to study visits from randomization to last visit.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey DESCHAMPS, PhD, Study Director — Kitozyme, Belgium; Xavier DEPLANQUE, MD, Principal Investigator — Clinical Nutrition Center Naturalpha, France
Locations (1):
- Clinical Nutrition Center Naturalpha (CNCN), Lille, France